CLINICAL TRIAL: NCT02688829
Title: The Initial Small-Scale Clinical Study of Rapamycin-Eluting Coronary Stent System of Microport (Firehawk)
Brief Title: The First-In-Man Pilot Study of Firehawk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Firehawk_FIM
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Results first posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-09

CONDITIONS: Coronary Heart Disease
Keywords: Sirolimus eluting stents; percutaneous coronary intervention; First in man
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment group (Experimental): Implantation of the rapamycin target-eluting coronary stent system (Firehawk)in patients with coronary heart disease.
  Interventions: Device: Rapamycin target-eluting Coronary Stent System

INTERVENTIONS:
Device: Rapamycin target-eluting Coronary Stent System — Implantation of the rapamycin-eluting coronary stent system
  Other Names: Firehawk

SUMMARY:
This is a small-scale pilot clinical study of the Rapamycin-Eluting Coronary Stent System of Microport for the first time to assess the preliminary safety and feasibility used in the human body. And provide evidence for subsequent large-scale, multi-center, randomized controlled clinical trials, then provide the basis for the formal application of the product in China.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age, males or non-pregnant females;
2. With silent ischemia evidence, patients with stable or unstable angina, or in patients with old myocardial infarction;
3. Total number of target lesion is 1;
4. Target lesion length ≤ 30mm (Visual); target lesion diameter between 2.25mm to 4.0mm;
5. Visual assessment of target lesion diameter stenosis ≥ 70%,TIMI blood flow≥1;
6. Each target lesion may be covered by a single stent;
7. Patients with indications for coronary artery bypass graft surgery;
8. To understand the purpose of testing, voluntary and informed consent, patients undergoing invasive imaging follow-up.

Exclusion Criteria:

1. Within 1 month of any acute myocardial infarction;
2. Chronic total occlusion (TIMI grade 0 flow before surgery), left main coronary artery disease, mouth lesions, multiple-vessel lesions, branch diameter ≥ 2.5mm bifurcation lesions and vascular lesions of the bridge;
3. Severe calcified lesions that cannot be successfully expanded and distorting lesions not suitable for stent delivery;
4. In-stent Restenosis lesions;
5. Intracoronary implantation of any branding stents within 1 year;
6. Severe congestive heart failure (NYHA class III and above) ,left ventricular ejection fraction or <40% (ultrasound or left ventricular angiography);
7. Preoperative renal function serum creatinine >2.0mg/DL;
8. Bleeding, active gastrointestinal ulcers, brain hemorrhage or subarachnoid hemorrhage and half year history of ischemic stroke, antiplatelet agents and would not allow an anticoagulant therapy contraindications patients undergoing antithrombotic therapy;
9. Aspirin, clopidogrel, heparin, contrast agent, poly lactic acid polymer and rapamycin allergies;
10. The patient's life expectancy is less than 12 months;
11. Top participated in other drug or medical device and does not meet the primary study endpoint in clinical trials time frame;
12. Researchers determine patient compliance is poor, unable to complete the study in accordance with the requirements;
13. Heart transplantation patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual); Study Completion 2015-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 21
Completed | 19
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Region of Enrollment [Count of Participants; unit: Participants]
  China | 21

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With MACE (Major Acute Cardiovascular Events)
Description: Count of Participants who have major acute cardiovascular events (MACE) in 1 month follow-up, MACE defined as the composite of cardiac death, myocardial infarction(Q and non-Q) and ischemia driven target lesion revascularization.
Time Frame: 1 month after stent implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
Participants | 0

2. Secondary Outcome: In-stent Late Lumen Loss
Description: In-stent late lumen loss (In-stent LLL) is defined as the difference between the post-procedure and 4 months follow-up in-stent minimal lumen diameter.
Time Frame: 4 months after stent implantation
Population: Angiographic follow-up at 4 months was obtained in 19 patients.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
mm | 0.13 (0.18)

3. Secondary Outcome: Count of Participants With MACE (Major Acute Cardiovascular Events)
Description: Count of Participants who have major acute cardiovascular events (MACE) in 4 months follow-up, MACE defined as the composite of cardiac death, myocardial infarction(Q and non-Q) and ischemia driven target lesion revascularization.
Time Frame: 4 month after stent implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
Participants | 0

4. Secondary Outcome: Percentage of In-stent Diameter Stenosis
Description: Percentage of in-stent diameter stenosis is calculated by the following fomula: (RVD-MLD)/RVD * 100%.
  RVD: Reference vessel diameter, represents the averaged diameter of the coronary assumed without atherosclerotic disease.
  MLD: Minimal luminal diameter, represents the smallest lumen diameter in the segment of interest.
Time Frame: 4 months after stent implantation
Population: Angiographic follow-up at 4 months was obtained in 19 patients.
Measure: Mean (Standard Deviation); unit: percentage of lumen diameter
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
percentage of lumen diameter | 13.4 (6.5)

5. Secondary Outcome: In-stent Late Lumen Loss
Description: In-stent late lumen loss (In-stent LLL) is defined as the difference between the post-procedure and 13 months follow-up in-stent minimal lumen diameter.
Time Frame: 13 month after stent implantation
Population: Angiographic follow-up at 13months was obtained in 19 patients.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
mm | 0.16 (0.07)

6. Secondary Outcome: Count of Participants With MACE (Major Acute Cardiovascular Events)
Description: Count of Participants who have major acute cardiovascular events (MACE) in 13 months follow-up, MACE defined as the composite of cardiac death, myocardial infarction(Q and non-Q) and ischemia driven target lesion revascularization.
Time Frame: 13 month after stent implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
Participants | 0

7. Secondary Outcome: Percentage of In-stent Diameter Stenosis
Description: as for outcome 4
Time Frame: 13 month after stent implantation
Population: Angiographic follow-up at 4 months was obtained in 19 patients.
Measure: Mean (Standard Deviation); unit: percentage of lumen diameter
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
percentage of lumen diameter | 12.9 (4.7)

ADVERSE EVENTS:
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 1/21
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=21)
TVR (Cardiac disorders) | 1 (1) — Target vessel revascularization, defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel.
Hemorrhagic stroke (Nervous system disorders) | 1 (1) — Hemorrhagic stroke is defined as a sudden onset of focal neurological deflicits due to cebral vascular bleeding that lasts more than 24 hours.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No